CLINICAL TRIAL: NCT07209215
Title: ULtra sensiTive ctDNA-Informed Management eArly-stage recTal cancEr (ULTIMATE)
Brief Title: ctDNA-Informed Management of Early-Stage Rectal Cancer
Acronym: ULTIMATE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC322; P30CA093373 (NIH)
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Rectal Adenocarcinoma; Rectal Cancer; Early-stage Rectal Cancer; Locally Advanced Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ctDNA informed management arm (Watch and Wait surveillance) (Experimental)
  Interventions: Drug: Signatera Genome ultra-sensitive ctDNA blood test + total neoadjuvant therapy (TNT)
- Post TNT SOC surgery arm (Experimental)
  Interventions: Drug: Signatera Genome ultra-sensitive ctDNA blood test + total neoadjuvant therapy (TNT)

INTERVENTIONS:
Drug: Signatera Genome ultra-sensitive ctDNA blood test + total neoadjuvant therapy (TNT) — Use of Signatera Genome ultra-sensitive ctDNA blood test post-total neoadjuvant therapy (TNT) for ctDNA-informed treatment management of early-stage rectal cancer.

SUMMARY:
This is a phase 2 pragmatic study to examine the utility of ctDNA-informed treatment management for participants with early-stage rectal cancer using the Signatera Genome assay. The primary aims are to 1) assess pathologic complete response (path CR) in the ctDNA informed management arm; 2) assess pathologic complete response (path CR) in the post total neoadjuvant therapy (TNT) standard of care (SOC) surgery arm; and 3) assess disease free survival (DFS) in the ctDNA informed management arm.

DETAILED DESCRIPTION:
Two cohorts of participants will be enrolled: Cohort A (participants appropriate for receiving TNT) and Cohort B (TNT already performed at UC Davis Health or externally). At Time A after TNT is completed and based on ctDNA assay results, the clinical decision will be made to put participants into one of two arms: the ctDNA informed management arm (Watchful Waiting [WW] surveillance) or the post TNT SOC surgery arm; participants will be monitored for ctDNA positivity for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Tumor tissue histologically confirming rectal adenocarcinoma that is available for Natera ctDNA assay.
* Cohort A only: Patients appropriate for receiving TNT including chemotherapy and chemoradiation.
* Cohort B only: TNT must have included at least 4 cycles of CAPEOX or 6 cycles of FOLFOX and at least 45 Gy in 25 fractions to the pelvis during chemoradiation.
* Patients ≥18 years of age at time of consent.
* Ability to understand and willingness to sign the informed consent form (ICF).
* Ability and stated willingness to adhere to the study visit schedule and protocol procedures/requirements.

Exclusion Criteria:

* Prior treatment for rectal cancer, except for cohort B.
* Evidence of distant metastatic disease on staging imaging (CT chest with abdominopelvic imaging by CT or MRI) within 8 weeks of enrollment.
* Patients on hemodialysis.
* Any condition that in the opinion of the investigator would interfere with the participant's safety or compliance while on trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pathCR) rate (ctDNA Informed Management Arm) | Up to 2 years after TNT
  Percent of participants with local regrowth within 2 years of total neoadjuvant therapy (TNT)
Pathologic complete response (pathCR) rate (Post TNT SOC Surgery Arm) | Up to 2 years after TNT
  Percent of participants with local regrowth within 2 years of TNT
Disease-free survival (DFS) rate (ctDNA Informed Management Arm) | Up to 2 years after TNT
  Median interval from first date of TNT to the first occurrence of locoregional failure, distant recurrence, a new invasive colorectal primary cancer.

SECONDARY OUTCOMES:
Frequency of local regrowth (ctDNA Informed Management Arm) | Up to 2 years after TNT
  Percentage of participants with local regrowth within 2 years of TNT

CONTACTS AND LOCATIONS:
Overall Officials: Ankit Sarin, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States